CLINICAL TRIAL: NCT01692015
Title: A Questionnaire Study on Diet and Hereditary Haemorrhagic Telangiectasia
Brief Title: Diet and Hereditary Haemorrhagic Telangiectasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CLS21
Record Dates: First submitted 2012-09-20; First posted 2012-09-25 (Estimated); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-09

CONDITIONS: Hereditary Haemorrhagic Telangiectasia (HHT)
Keywords: Hereditary Haemorrhagic Telangiectasia; Nose bleeding; Iron supplements
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Hematologic Tests; Blood Cell Count; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet and nosebleed questionnaire (Experimental): Participants will only be required to fill in two paper questionnaires, one on dietary history, and one on nosebleed severity.
  Interventions: Other: Questionnaire on dietary history; Other: Questionnaire on nosebleed severity
- Weighed food diary arm (Experimental): Participants will be required to weigh their food for one week to generate a food dairy, and have a single blood test, in addition to filling in the two paper questionnaires, one on dietary history, and one on nosebleed severity.
  Interventions: Other: Questionnaire on dietary history; Other: Questionnaire on nosebleed severity; Other: One week food diary generated by weighing foods; Procedure: Blood tests for full blood count, albumin, and indices of nutritional status

INTERVENTIONS:
Other: Questionnaire on dietary history
Other: Questionnaire on nosebleed severity
Other: One week food diary generated by weighing foods
  Arms: Weighed food diary arm
Procedure: Blood tests for full blood count, albumin, and indices of nutritional status
  Arms: Weighed food diary arm

SUMMARY:
Hereditary Haemorrhagic Telangiectasia (HHT) affects 1 in 5,000 people. The purpose of this study is to provide data regarding the diet and nosebleed frequency using a questionnaire.

This will be filled in by people with HHT.

The questionnaire has been designed in paper format.

DETAILED DESCRIPTION:
Hereditary Haemorrhagic Telangiectasia (HHT) affects 1 in 5,000 people, usually causing nosebleeds, skin blood spots, and/or anaemia as a result of bleeding from the nose or gut. The majority of people with HHT also have abnormal blood vessels (arteriovenous malformations) in internal organs such as the lungs, liver and brain. Management of this multisystem disorder is highly challenging.

The Lead Applicant has spent 20 years working on this rare disease, and identified multiple areas where more evidence is required to assist clinicians and patients with this lifelong condition. A particular issue is whether the diet influences HHT or its complications in any way.

In this study, people will fill in two questionnaires, one giving details of their diet, and another details of their nosebleeds. They will also be asked to consider participating in an accessory study arm which includes weighing food for one week and providing a food diary, in addition to having a single set of blood test.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of hereditary Haemorrhagic Telangiectasia (HHT)

Exclusion Criteria:

* Unable to provide informed consent
* Presence of another major organ disorder that may affect nutritional status, such as inflammatory bowel disease, or celiac disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire L Shovlin, PhD FRCP, Principal Investigator — Imperial College London
Locations (1):
- HHTIC London, Hammersmith Hospital, Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finnamore H, Le Couteur J, Hickson M, Busbridge M, Whelan K, Shovlin CL. Hemorrhage-adjusted iron requirements, hematinics and hepcidin define hereditary hemorrhagic telangiectasia as a model of hemorrhagic iron deficiency. PLoS One. 2013 Oct 16;8(10):e76516. doi: 10.1371/journal.pone.0076516. eCollection 2013. PMID 24146883
- [Result] Finnamore HE, Whelan K, Hickson M, Shovlin CL. Top dietary iron sources in the UK. Br J Gen Pract. 2014 Apr;64(621):172-3. doi: 10.3399/bjgp14X677761. No abstract available. PMID 24686867
- [Result] Chamali B, Finnamore H, Manning R, Laffan MA, Hickson M, Whelan K, Shovlin CL. Dietary supplement use and nosebleeds in hereditary haemorrhagic telangiectasia - an observational study. Intractable Rare Dis Res. 2016 May;5(2):109-13. doi: 10.5582/irdr.2016.01019. PMID 27195194
- [Result] Finnamore H, Silva BM, Hickson BM, Whelan K, Shovlin CL. 7-day weighed food diaries suggest patients with hereditary hemorrhagic telangiectasia may spontaneously modify their diet to avoid nosebleed precipitants. Orphanet J Rare Dis. 2017 Mar 28;12(1):60. doi: 10.1186/s13023-017-0576-6. PMID 28347346

RESULTS

PARTICIPANT FLOW:
Groups:
- Hereditary Hemorrhagic Telangiectasia (HHT): Patients with hereditary hemorrhagic telangiectasia (HHT)
Period: Overall Study
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 55 [20 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieving Personal Recommended Intake of Iron
Description: Dietary food item iron content assessed by the European Prospective Investigation into Cancer and Nutrition (EPIC) food frequency questionnaire. This method has been validated against the gold standard for dietary assessment, a 7-day weighed food diary. Questions are asked about consumption of 130 major food items over the previous year, requiring participants to indicate the frequency of consumption, and to provide details about the methods of cooking, type of produce, and use of dietary supplements. The EPIC FFQ has been widely validated in a number of studies and is deemed an adequate assessment tool to assess dietary intake.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
Number analyzed (Participants) | 50
Participants | 43

2. Primary Outcome: Nosebleed Severity
Description: Nosebleeds were quantified using the validated Epistaxis Severity Score (ESS). The six questions provide an objective measure of nosebleeds: three relate to different characteristics of typical nosebleeds within the previous three months (frequency, duration and intensity (gushing/pouring or not)), three to medical attention, anemia and transfusion requirements. The final ESS score ranges from 0-10, where a higher score equates to greater blood losses.
Time Frame: 3 months
Measure: Median (Full Range); unit: units
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
Number analyzed (Participants) | 50
units | 4.4 [0 to 9.1]

3. Primary Outcome: Number of Participants That Achieving the Hemorrhage Adjusted Iron Requirement (HAIR)
Description: The hemorrhage-adjusted iron requirement (HAIR) was calculated as the sum of the normal recommended dietary iron intake, and requirements to compensate for non-menstrual blood losses.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
Number analyzed (Participants) | 50
Participants | 10

4. Other Pre Specified Outcome: Number of Participants That Ingested Chocolate
Description: Chocolate can precipitate nosebleeds Food items intake assessed by 7-day weighed food diary
Time Frame: 3 months
Population: 25 participants were filled up the 7-day weighed food diary
Measure: Count of Participants; unit: Participants
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
Number analyzed (Participants) | 25
Participants | 14

5. Other Pre Specified Outcome: Number of Participants That Ingested Bread
Description: Bread not precipitate nosebleeds Food items intake assessed by 7-day weighed food diary
Time Frame: 3 months
Population: 25 participants were filled up the 7-day weighed food diary
Measure: Count of Participants; unit: Participants
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Hereditary Hemorrhagic Telangiectasia (HHT)
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes